CLINICAL TRIAL: NCT02120742
Title: The Impact Of Text Message (SMS) Reminders On Helmet Use Among Motorcycle Drivers In Dar Es Salaam, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amend (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D14103
Record Dates: First submitted 2014-04-19; First posted 2014-04-23 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Road Traffic Injury Prevention; Helmet Use; mHealth Intervention
Keywords: Road traffic injury prevention; Helmet use; mHealth intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Social Norming (Experimental): The first group will receive SMS message reminders framed as social norming (ie "Most of your peers wear helmets").
  Interventions: Behavioral: SMS message reminder
- Fear Appeal (Experimental): The second group will receive SMS message reminders framed as fear appeals (ie "Not wearing your helmet increases your chance of dying in an accident").
  Interventions: Behavioral: SMS message reminder
- Control (Placebo Comparator): The third group will act as the control and receive texts that relate to general road safety, but not helmet use.
  Interventions: Behavioral: SMS message reminder

INTERVENTIONS:
Behavioral: SMS message reminder — SMS texts will be delivered to study participants over a 6-week period.

SUMMARY:
This study seeks to evaluate the impact of a text-message (SMS) program delivered to motorcycle drivers in Dar es Salaam, Tanzania. The SMS program, delivered by nonprofit Amend, sends daily reminders to motorcycle drivers to remind them to wear their helmets. In this study, the investigators will conduct a randomized controlled trial to see if this program leads to increased helmet use over time. The investigators will recruit between 350-400 motorcycle drivers to receive the text program. The investigators will obtain each of their cell phone numbers, and the participants will be split into three groups. The first group will receive reminders framed as social norming (ie "Most of your peers wear helmets"). The second group will receive reminders framed as fear appeals (ie "Not wearing your helmet increases your chance of dying in an accident"). The third group will act as the control and receive texts that relate to general road safety, but not helmet use. All groups will receive the same general road safety information being delivered to the control arm. The purpose of sending different types of reminders is to assess which type of messages are more likely to cause a motorcycle driver to regularly wear their helmet. The investigators will survey the participants at the initiation of the study and after weeks 3 and 6 during the study, asking about their helmet use. This will be a short survey, and any personal information gathered during the study (ie, phone numbers), will be securely stored so as to protect their privacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Must own a cell phone with text-message features
* Must demonstrate ability to retrieve and read text-messages
* Must have access to a helmet.

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Self-reported adherence to helmet use | Midpoint of study (3 weeks)
  The primary outcome of the study will be self-reported adherence to helmet use as measured by the proportion of participants who wear their helmet on all trips
Self-reported adherence to helmet use | Endpoint of study (6 weeks)
  The primary outcome of the study will be self-reported adherence to helmet use as measured by the proportion of participants who wear their helmet on all trips

SECONDARY OUTCOMES:
Attitude change | 6 weeks
  A secondary outcome will be participants' attitudes toward helmet use and the SMS reminder platform, as measured by an open-ended survey at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Upanga West, Tanzania

REFERENCES:
- [Derived] Campbell B, Heitner J, Amos Mwelelo P, Fogel A, Mujumdar V, Adams LV, Boniface R, Su Y. Impact of SMS Text Messaging Reminders on Helmet Use Among Motorcycle Drivers in Dar es Salaam, Tanzania: Randomized Controlled Trial. J Med Internet Res. 2022 Apr 7;24(4):e27387. doi: 10.2196/27387. PMID 35389364